CLINICAL TRIAL: NCT00971984
Title: Demographic, Clinical and Laboratory Characteristics of Children With Alpha Thalassemia in Northern Israel
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Dr Koren Ariel, Head of Pediatric Hematology Unit and Pediatric Dpt B, HaEmek Medical Center, Israel
Other Study IDs: 0074-09-EMC
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Thalassemia Alpha; Hemolytic Anemia
MeSH Terms: conditions — alpha-Thalassemia; Anemia, Hemolytic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Alpha thalassemia patients: Patients diagnosed with alpha thalassemia mutations and anemia
  Interventions: Other: Medical records summary

INTERVENTIONS:
Other: Medical records summary — Summary of Medical files and laboratory results.

SUMMARY:
The study intends to summarize the clinical and laboratory characteristics of children with hemolytic anemia diagnosed as having alpha thalassemia mutations.

DETAILED DESCRIPTION:
Fifty children and adolescents diagnosed as having alpha thalassemia will be studied, the clinical characteristics and hematology analysis will be summarized.

ELIGIBILITY:
Inclusion Criteria:

* All the patients that were studied at the pediatric hematology unit ant the Ha'Emek Medical Center

Exclusion Criteria:

* None

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A group of 50 children that underwent workup due to hemolytic anemia and were further diagnosis as suffering from clinical alpha thalassemia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2009-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Analysis of the Demographic, Clinical and Laboratory Characteristics of Children With Alpha Thalassemia | One year
  Analysis of the Demographic, Clinical and Laboratory Characteristics of Children With Alpha Thalassemia

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Hematology Unit and Pediatric Dpt B - HaEmek Medical Center, Afula, Israel